CLINICAL TRIAL: NCT05083494
Title: Real-time Monitoring of Concentration and Size Variations of Circulating Plasma Free DNA to Predict Early Response to Immunotherapies in Patients With Different Types of Cancer.
Acronym: SCHISM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-048
Record Dates: First submitted 2021-10-06; First posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Melanoma
- clear cell renal cancer
- Urothelial Carcinoma of the bladder
- squamous cell carcinomas of the head and neck
- non-small cell lung cancer

SUMMARY:
Immunotherapy, which can be represented by the immune checkpoint blockade, is a milestone in the progress of the ongoing struggle against cancer. However, the emergence of unexpected tumor response patterns, such as pseudo-progression or hyper-progression, might complicate the management of patients receiving these immune checkpoint inhibitors. A reliable standardized biomarker that can be used in clinical practice for predicting response to treatment, monitoring tumor evolution and evaluating treatment efficacy has not yet been established.

The general aim of this study is to assess the interest of the plasmatic free circulating DNA (cfDNA) on the clinical response for patients with different types of cancer treated with immunotherapies. The primary objective is to assess the performance of the plasmatic free circulating DNA using the estimation of the receiver operating characteristic (ROC) curve and calculation of the area under the curve (AUC) on the response rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients starting anti-PD1 immunotherapy as part of marketing authorization alone or in combination (melanoma, clear cell renal cancer, urothelial carcinomas of the bladder, squamous cell carcinomas of the head and neck and non-small cell lung cancer).
* No contraindications to immunotherapy
* Non-pregnant patient
* Patient not opposed to participation in this study

Exclusion Criteria:

* HIV seropositivity
* Patient with psychiatric or other conditions that may compromise his or her ability to give non opposition or to follow study procedures

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients starting a cancer treatment, as part of marketing treatment (alone or in combination) in five type of cancer (melanoma, clear cell renal cancer, urothelial carcinomas of the bladder, squamous cell carcinomas of the head and neck and non-small cell lung cancer).
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2021-04-09 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Interest of the plasmatic free circulating DNA (cfDNA) | At first evaluation, then 1 administration over 2 for 1 year then at 18 months and an additional sample will be taken at the time of recurrence
  The primary objective is to assess the performance of the plasmatic free circulating DNA using the estimation of the receiver operating characteristic (ROC) curve and calculation of the area under the curve (AUC) on the response rate

CONTACTS AND LOCATIONS:
Locations (1):
- APHM, Marseille, France